CLINICAL TRIAL: NCT02346747
Title: A Randomized, Double-Blind, Placebo-Controlled Phase 2 Trial of Vigil Engineered Autologous Tumor Cell Immunotherapy in Subjects With Stage IIIb-IV Ovarian Cancer in Clinical Complete Response Following Surgery and Primary Chemotherapy
Brief Title: A Trial of Vigil for Participants With Ovarian Cancer
Acronym: VITAL
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Gradalis, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CL-PTL-119
Record Dates: First submitted 2015-01-21; First posted 2015-01-27 (Estimated); Last update posted 2025-10-29 (Actual); Status verified 2025-10

CONDITIONS: Ovarian Cancer; Ovarian Neoplasms
Keywords: Stage III; Stage IV; Ovarian Cancer; Maintenance; Immunotherapy; primary peritoneal cancer; fallopian tube cancer; endometrioid ovarian cancer; high-grade serous ovarian cancer
MeSH Terms: conditions — Ovarian Neoplasms; Fallopian Tube Neoplasms | interventions — FANG vaccine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Group A (Active Comparator): Vigil immunotherapy will be administered at a concentration of 1.0 x 10e7 cells/dose given via intradermal injection every 4 weeks for a minimum of 4 and a maximum of 6 administrations as determined by the number of doses manufactured and as long as the subject is clinically stable and recurrence free.
  Interventions: Biological: Vigil
- Group B (Placebo Comparator): Placebo will be administered via intradermal injection every 4 weeks for a minimum of 4 and a maximum of 6 administrations as determined by the number of doses manufactured and as long as the subject is clinically stable and recurrence free.
  Interventions: Other: Placebo

INTERVENTIONS:
Biological: Vigil — The bi-shRNAfurin and GMCSF Augmented Autologous Tumor Cell Vaccine, Vigil is made up of irradiated autologous tumor cells which have been electroporated ex vivo with the Vigil plasmid designed to suppress expression of both the TGFβ1 and TGFβ2 proteins while simultaneously expressing rhGMCSF protein.
  Other Names: bi-shRNAfurin and GMCSF Autologous Tumor Cell Immunotherapy; FANG vaccine
  Arms: Group A
Other: Placebo — To maintain placebo effect and eliminate bias due to volumetric differences, the number of Vigil doses manufactured from harvested tissue (except if below 4) will be used to guide manufacture of the same number of doses of placebo for each subject. Placebo will consist of "freeze" media [10% DMSO (dimethyl sulfoxide; Cryoserv USP; Mylan Institutional USP), 1% Human Serum Albumin (ABO Pharmaceuticals) in Plasma-Lyte A, pH 7.4 (Baxter)]. Depending upon randomization assignment, placebo or Vigil will be delivered in identical vials and drawn up in 'covered' syringes for intradermal injection.
  Arms: Group B

SUMMARY:
The goal of this clinical trial is to compare participants with ovarian, fallopian tube or primary peritoneal cancer when treated with investigational product (Vigil) compared to placebo. The main question it aims to answer is "Will participants who receive treatment with Vigil have a longer time to disease recurrence versus the participants that were not given Vigil?"

DETAILED DESCRIPTION:
This is a multicenter, randomized, double-blind, placebo-controlled, Phase 2 study of maintenance Vigil Ovarian (gemogenovatucel-T) engineered autologous tumor cells (EATC) in women with Stage IIIb, IIIc or IV high-grade papillary serous/ clear cell / endometrioid ovarian, fallopian tube or primary peritoneal cancer. Subjects will have had a minimum of 4 and a maximum of 12 doses of Vigil prepared and stored from ovarian tumor cells obtained at the time of primary surgical debulking or initial diagnostic / evaluative laparoscopy (tissue for immunotherapy manufacture must be procured prior to initiation of neoadjuvant chemotherapy). An equal number of placebo doses will be manufactured. Subjects eligible for randomization will have achieved a clinically defined complete response following primary surgery and adjuvant chemotherapy. Clinical complete response (cCR) is defined as no evidence of maligancy on chest x-ray and CT scan or MRI of the abdomen and pelvis, CA-125 antigen level ≤ units/mL, and no findings on physical examination or symptoms suggestive of active cancer.

Investigational treatment must start no less than 3 weeks and no more than 8 weeks following completion of chemotherapy.

Approximately 86 subjects will be randomized 1:1 to to Group A (Vigil 1.0 X 10e7 cells/injection) or Group B (placebo). Randomization will be stratified by (i) extent of surgical cytoreduction (complete/microscopic versus macroscopic residual disease) and (ii) neoadjuvant versus adjuvant chemotherapy. Participants will receive Vigil or placebo by intradermal injection once a month for at least 4 and up to a maximum of 6 doses determined by the number of doses of Vigil manufactured for that subject.

Participants will be managed in an outpatient setting. Image assessment with chest x-ray and CT scan or MRI of the abdomen and pelvis will be completed every 3 months in Years 1-3, then every 6 months in Years 4 and 5 and yearly through Year 10. At the time the participant recurs, the participant will enter long term follow-up for survival status and post treatment therapies received.

ELIGIBILITY:
Inclusion Criteria

Subjects will be eligible for tissue procurement for the Vigil manufacturing process if they meet all of the following criteria:

1. Presumptive Stage IIIb, IIIc or IV high-grade papillary serous/clear cell/endometrioid ovarian, fallopian tube or primary peritoneal cancer.
2. No chemotherapy prior or investigational agents prior to tissue acquisition for Vigil manufacture.
3. No other malignancy (excluding surgically cured nonmelanoma carcinomas of the skin and carcinoma in situ cervix) unless in remission for ≥ 2 years.
4. Anticipated availability of a cumulative mass of ~30 grams tissue ("golf-ball" size or approximately 3cm disease on CT scan) at time of diagnostic laparoscopy or primary surgical debulking. Infiltrating lumen (bowel, fallopian tube, urethra) tissue should not be used as Vigil immunotherapy material to minimize risk of bacterial contamination.
5. ECOG performance status (PS) 0-2 prior to diagnostic laparoscopy or debulking laparotomy.
6. No prior history of hypersensitivity reactions (HSR) with taxanes or platinums.
7. No prior history of allergies or sensitivities to gentamicin.
8. Female, 18 years of age or older.
9. Ability to understand and the willingness to sign a written informed consent document for tissue harvest.

Subjects will be registered in this study if they meet all of the following inclusion criteria:

1. Histologically confirmed Stage IIIb, IIIc or IV high-grade papillary serous/clear cell/endometrioid ovarian, fallopian tube or primary peritoneal.
2. Completion of primary surgical debulking including hysterectomy and bilateral salpingo oophorectomy, and at least 5 but no more than 8 cycles of platinum / taxane adjuvant chemotherapy or chemotherapy as per Category 1 recommendations of the NCCN guidelines, including 5-8 cycles adjuvant intraperitoneal + intravenous (IP/IV) chemotherapy, or 5-8 cycles of intravenous chemotherapy divided and administered as neoadjuvant and adjuvant therapy flanking primary debulking surgery.
3. Clinically defined complete response (cCR) following completion of primary surgical debulking and eligible chemotherapy. cCR defined as no evidence of malignancy on chest x-ray (CT scan is acceptable) and CT scan or MRI of the abdomen and pelvis, normal physical examination, CA-125 antigen level ≤ 35 U/ml (assessed ≥ 2 weeks following removal of catheter in subjects receiving intraperitoneal/intravenous chemotherapy) and no findings on physical examination or symptoms suggestive of active cancer.
4. Subjects must have initiated adjuvant chemotherapy no more than 8 weeks following primary debulking surgery.
5. Successful manufacturing of at least 4 doses (vials) of Vigil and placebo.
6. Recovered from all clinically relevant toxicities related to prior therapy (including neuropathy ≤Grade 2).
7. ECOG performance status (PS) 0-1.
8. Normal organ and marrow function as defined below: Absolute granulocyte count ≥ 1,500/mm^3, Absolute lymphocyte count ≥ 500/mm^3, Platelets ≥ 75,000/mm^3, Total bilirubin ≤ 2 mg/dL, AST(SGOT)/ALT(SGPT)≤ 2x institutional upper limit of normal, Creatinine < 1.5 mg/dL
9. Ability to understand and the willingness to sign a written informed protocol specific consent.

Exclusion Criteria:

Subjects will be excluded from this study if they meet any of the following criteria (at the time of tissue procurement or at randomization):

1. Surgery involving general anesthesia, radiotherapy, immunotherapy, or investigational agents within 4 weeks prior to randomization.
2. Histologically confirmed papillary serous adenocarcinoma of the uterus or disease involving myometrium/endometrium.
3. Systemic immunosuppressive therapy within 14 days of randomization.
4. Subjects requiring chronic steroid or immunosuppressive regimens are excluded except inhaled / intranasal steroids and short term systemic steroids <30 days duration and ≤0.25 mg/kg prednisone-equivalent per day are allowed.
5. Congestive heart failure (NYHA Class II, III, or IV), unstable angina, ventricular or hemodynamically significant atrial arrhythmia, or cardiovascular disease such as stroke or myocardial infarction (current or within the past 6 months).
6. Psychiatric illness/social situations that would limit compliance with study requirements.
7. Subjects with history of brain metastases.
8. Subjects with known HIV or chronic Hepatitis B or C infection.
9. Prior solid organ or bone marrow transplant.
10. History of or active autoimmune disease (e.g., autoimmune neutropenia, thrombocytopenia, or hemolytic anemia, systemic lupus erythematosus, Sjogren's syndrome, scleroderma, myasthenia gravis, Goodpasture's syndrome, Addison's disease, Hashimoto's thyroiditis, or Graves disease). Persons with vitiligo are not excluded. Diabetics are not excluded if the condition is well controlled.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 92 (Actual)
Dates: Start 2015-02 (Actual); Primary Completion 2028-12 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Recurrence Free Survival (RFS) | Time from randomization date to either the date of first recurrence or the date of death if the participant dies prior to recurrence, assessed up to 10 years.
  Disease recurrence will be evaluated using the Response Evaluation Criteria in Solid Tumors (RECIST) Version 1.1 by local and central radiology. RFS is defined as the time from randomization or from surgery/procurement to the event of disease recurrence/progression or death due to any cause.

SECONDARY OUTCOMES:
Overall survival (OS) | OS will be evaluated from time of randomization until date of death can be obtained, assessed up to 10 years.
  OS is defined as the time from randomization to date of death due to any cause.

CONTACTS AND LOCATIONS:
Overall Officials: John Nemunaitis, MD, Study Director — Gradalis, Inc.
Locations (26):
- United States (26):
  - University of South Alabama Mitchell Cancer Institute, Mobile, Alabama
  - Southern California Permanente Medical Group, Irvine, California
  - Palo Alto Foundation Medical Group, San Francisco, California
  - University Of Miami Sylvester Comprehensive Cancer Center, Miami, Florida
  - Moffitt Cancer Center, Tampa, Florida
  - Florida Cancer Specialists, West Palm Beach, Florida
  - Georgia Cancer Center at Augusta University, Augusta, Georgia
  - University Of Kentucky Markey Cancer Center, Lexington, Kentucky
  - Maine Medical Center: MMP Women's Health, Scarborough, Maine
  - Dana Farber Cancer Institute: Gynecologic Oncology, Boston, Massachusetts
  - Henry Ford Health System, Detroit, Michigan
  - Billings Clinic, Billings, Montana
  - Nebraska Methodist Hospital, Omaha, Nebraska
  - Dartmouth-Hitchcock Medical Center/Norris Cotton Cancer Center, Lebanon, New Hampshire
  - University of New Mexico Cancer Center, Albuquerque, New Mexico
  - Duke University Medical Center, Department of Medicine - Oncology, Durham, North Carolina
  - Barrett Cancer Center University of Cincinnati Medical Center, Cincinnati, Ohio
  - Stephenson Cancer Center at University of Oklahoma, Oklahoma City, Oklahoma
  - AMD Asplundh Cancer Pavilion, Abington, Pennsylvania
  - St. Luke's Health Network, Bethlehem, Pennsylvania
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - Prisma Health Cancer Institute, Greenville, South Carolina
  - Mary Crowley Cancer Research Centers, Dallas, Texas
  - University of Texas Southwestern Medical Center, Dallas, Texas
  - Cancer Care Northwest, Spokane, Washington
  - Franciscan Research Center, Tacoma, Washington

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Senzer N, Barve M, Kuhn J, Melnyk A, Beitsch P, Lazar M, Lifshitz S, Magee M, Oh J, Mill SW, Bedell C, Higgs C, Kumar P, Yu Y, Norvell F, Phalon C, Taquet N, Rao DD, Wang Z, Jay CM, Pappen BO, Wallraven G, Brunicardi FC, Shanahan DM, Maples PB, Nemunaitis J. Phase I trial of "bi-shRNAi(furin)/GMCSF DNA/autologous tumor cell" vaccine (FANG) in advanced cancer. Mol Ther. 2012 Mar;20(3):679-86. doi: 10.1038/mt.2011.269. Epub 2011 Dec 20. PMID 22186789
- [Background] Nemunaitis J, Barve M, Orr D, Kuhn J, Magee M, Lamont J, Bedell C, Wallraven G, Pappen BO, Roth A, Horvath S, Nemunaitis D, Kumar P, Maples PB, Senzer N. Summary of bi-shRNA/GM-CSF augmented autologous tumor cell immunotherapy (FANG) in advanced cancer of the liver. Oncology. 2014;87(1):21-9. doi: 10.1159/000360993. Epub 2014 Jun 25. PMID 24968881
- [Background] Senzer N, Barve M, Nemunaitis J, Kuhn J, Melnyk A, et al. (2013) Long Term Follow Up: Phase I Trial of "Bi-Shrnafurin/GMCSF DNA/Autologous Tumor Cell" Immunotherapy (FANG™) in Advanced Cancer. J Vaccines Vaccin 4:209. doi: 10.4172/2157-7560.1000209
- [Background] Ghisoli M, Barve M, Mennel R, Lenarsky C, Horvath S, Wallraven G, Pappen BO, Whiting S, Rao D, Senzer N, Nemunaitis J. Three-year Follow up of GMCSF/bi-shRNA(furin) DNA-transfected Autologous Tumor Immunotherapy (Vigil) in Metastatic Advanced Ewing's Sarcoma. Mol Ther. 2016 Aug;24(8):1478-83. doi: 10.1038/mt.2016.86. Epub 2016 Apr 25. PMID 27109631
- [Background] Ghisoli M, Barve M, Schneider R, Mennel R, Lenarsky C, Wallraven G, Pappen BO, LaNoue J, Kumar P, Nemunaitis D, Roth A, Nemunaitis J, Whiting S, Senzer N, Fletcher FA, Nemunaitis J. Pilot Trial of FANG Immunotherapy in Ewing's Sarcoma. Mol Ther. 2015 Jun;23(6):1103-1109. doi: 10.1038/mt.2015.43. Epub 2015 Mar 19. PMID 25917459
- [Background] Oh J, Barve M, Senzer N, Aaron P, Manning L, Wallraven G, Bognar E, Stanbery L, Horvath S, Manley M, Nemunaitis J, Walter A, Rocconi RP. Long-term follow-up of Phase 2A trial results involving advanced ovarian cancer patients treated with Vigil(R) in frontline maintenance. Gynecol Oncol Rep. 2020 Sep 17;34:100648. doi: 10.1016/j.gore.2020.100648. eCollection 2020 Nov. No abstract available. PMID 33364285
- [Result] Rocconi RP, Grosen EA, Ghamande SA, Chan JK, Barve MA, Oh J, Tewari D, Morris PC, Stevens EE, Bottsford-Miller JN, Tang M, Aaron P, Stanbery L, Horvath S, Wallraven G, Bognar E, Manning L, Nemunaitis J, Shanahan D, Slomovitz BM, Herzog TJ, Monk BJ, Coleman RL. Gemogenovatucel-T (Vigil) immunotherapy as maintenance in frontline stage III/IV ovarian cancer (VITAL): a randomised, double-blind, placebo-controlled, phase 2b trial. Lancet Oncol. 2020 Dec;21(12):1661-1672. doi: 10.1016/S1470-2045(20)30533-7. PMID 33271095
- [Result] Rocconi RP, Monk BJ, Walter A, Herzog TJ, Galanis E, Manning L, Bognar E, Wallraven G, Stanbery L, Aaron P, Senzer N, Coleman RL, Nemunaitis J. Gemogenovatucel-T (Vigil) immunotherapy demonstrates clinical benefit in homologous recombination proficient (HRP) ovarian cancer. Gynecol Oncol. 2021 Jun;161(3):676-680. doi: 10.1016/j.ygyno.2021.03.009. Epub 2021 Mar 11. PMID 33715892